CLINICAL TRIAL: NCT04858828
Title: Investigation on Molecular Markers Associated With the Clinical Efficacy of Immunotherapy Combined With Chemotherapy in the First-line Treatment of Patients With Advanced Non-small-cell Lung Cancer
Brief Title: Investigation on Predictive Molecular Markers of Efficacy for Front-line Immunochemotherapy in Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Chief physician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: CROC2101
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a real-world exploratory study aiming to explore potential molecular markers detectable at baseline that can enable the prediction of clinical efficacy of front-line immunotherapy combined with chemotherapy in advanced non-small cell lung cancer (NSCLC). This study aims to include a total of 200 treatment-naïve patients initially diagnosed with advanced NSCLC. Paired tissue and blood samples collected from all patients before the start of immunochemotherapy treatment (baseline) will be analyzed. The patient samples will be submitted for molecular analysis, including next-generation sequencing (NGS)-based gene expression profiling (GEP) and inflammation-related T-cell receptor (TCR) repertoire profiling. The molecular assay results will include but will not be limited to tumor mutation burden (TMB), microsatellite instability (MSI) status, DNA damage repair (DDR)-related gene mutation status, and programmed death-ligand 1 (PD-L1) expression level. Patients will be followed-up for treatment responses until radiological confirmation of disease progression to first-line immunochemotherapy. The molecular assay results will then be analyzed with clinical data including objective responses and progression-free survival outcomes, among others, to identify molecular markers at baseline that are associated with clinical efficacy of immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are clinically diagnosed with stage IV NSCLC;
2. Patients who submitted samples for molecular testing using the OncoScreen Plus panel and PD-L1 (22C3) immunohistochemistry test at baseline;
3. Patients with negative results for sensitizing mutations for 6 genes, including EGFR, ALK, ROS1, BRAF, MET exon 14 skipping, and RET;
4. Patients without contraindications for immunotherapy;
5. Patients who are 18 years or older at the time of signing the informed consent form;
6. Patients with life expectancy of at least 12 weeks;
7. Patients with ECOG score of 0 or 1;
8. Patients with adequate organ function defined by the following criteria:

   1. Absolute neutrophil count ≥ 1.5109/L;
   2. Platelets ≥ 90109/L;
   3. Hemoglobin ≥ 9.0g/dL;
   4. Albumin levels ≥2.8 g/L;
   5. Total serum bilirubin ≤ 1.5 the upper limit of normal (ULN); for patients with liver metastases, total bilirubin ≤ 2 ULN;
   6. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN; for patients with liver metastases, ALT and AST ≤ 5ULN;
   7. Serum creatinine ≤ 1.5 ULN;
   8. International normalized ratio (INR) or plasma prothrombin time (PT) ≤1.5ULN.

Exclusion Criteria:

1. Patients with other concurrent tumors;
2. Patients with other concurrent medical conditions that may affect their follow-up and short-term survival;
3. Patients with any history of immunotherapy;
4. Patients with any history of chemotherapy, radiotherapy or other anti-tumor treatments;
5. Patients with heart function classified as New York Heart Association (NYHA) class III or IV;
6. Patients with peripheral nerve disease;
7. Patients with confirmed hearing loss;
8. Patients with other conditions deemed unsuitable for enrollment by the researchers.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC eligible for front-line treatment of immunotherapy combined with chemotherapy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Investigation on molecular markers associated with the clinical efficacy of immunotherapy combined with chemotherapy in the first-line treatment of patients with advanced non-small-cell lung cancer | June 2021 - March 2024
  Next-generation sequencing (NGS)-based gene expression profiling (GEP) and inflammation-related T-cell receptor (TCR) repertoire profiling. The molecular assay results will include but will not be limited to tumor mutation burden (TMB), microsatellite instability (MSI) status, DNA damage repair (DDR)-related gene mutation status, and programmed death-ligand 1 (PD-L1) expression level.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China